CLINICAL TRIAL: NCT04674228
Title: Review of Post-Study Clinical Endoscopy Reports in Follow Up to MAY2016-07-01 Weekly Erlotinib for Familial Adenomatous Polyposis
Brief Title: Review of Post-Study Clinical Endoscopy Reports in Follow Up to MAY2016-07-01
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: NCI-2020-13238; NCI-2020-13238 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); N01-CN-2012-00042; MAY2016-07-01F (Other: Mayo Clinic in Rochester); MAY2016-07-01F (Other: DCP); N01CN00042 (NIH); P30CA015083 (NIH)
Record Dates: First submitted 2020-12-17; First posted 2020-12-19 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Familial Adenomatous Polyposis
MeSH Terms: conditions — Adenomatous Polyposis Coli

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational (medical record review): Patients who participated in MAY2016-07-01 undergo review of medical records.
  Interventions: Other: Electronic Health Record Review

INTERVENTIONS:
Other: Electronic Health Record Review — Review of medical records

SUMMARY:
This study reviews post study clinical endoscopy reports in follow up to patients who participated in MAY2016-07-01 with weekly erlotinib for familial adenomatous polyposis. Reviewing follow up medical records may help researchers examine the extent of rapid progression of familiar adenomatous polyposis disease burden after discontinuation of weekly erlotinib.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To review clinical endoscopy reports, pathology reports, and other medical records related to standard-of-care endoscopic evaluations for all participants in the parent study, MAY2016-07-01, to determine the extent of reports of rapid progression of recurrent polyps after completion intervention and follow up under the parent protocol.

OUTLINE:

Patients who participated in MAY2016-07-01 undergo review of medical records.

ELIGIBILITY:
Inclusion Criteria:

* MAY2016-07-01 study participants for whom medical records are available and accessible

Exclusion Criteria:

* MAY2016-07-01 study participants who have opted out of medical records reviews or for whom consent for medical record review cannot be confirmed/documented

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants in MAY2016-07-01 Phase II Trial of Weekly Erlotinib Dosing to Reduce Duodenal Polyp Burden Associated with Familial Adenomatous Polyposis
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2021-05-07 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2022-05-17 (Actual)

PRIMARY OUTCOMES:
Number of study participants exhibiting clinically significant progression of duodenal neoplasia after completion of study drug | At completion of study
  Will be assessed by endoscopy.
Number of participants who underwent surgical resection | At completion of study
  Will determine the number of participants who underwent surgical resection for management of advanced upper gastrointestinal (GI) neoplasia/cancer between the date of completion of intervention and 2/28/2021.
Number of participants who required endoscopic resection of advanced upper gastrointestinal (GI) neoplasms | At completion of study

SECONDARY OUTCOMES:
Number of participants with evidence of progression of upper GI disease | At completion of study
  Will be calculated by increase in Spigelman stage.

CONTACTS AND LOCATIONS:
Overall Officials: Niloy J Samadder, Principal Investigator — Mayo Clinic in Rochester
Locations (2):
- United States (2):
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - M D Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm